CLINICAL TRIAL: NCT00377754
Title: A Prospective Study of Dengue Virus Infections During Infancy to Define Correlates of Protective Immunity
Brief Title: Prospective Study of Infant Dengue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0013
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-10

CONDITIONS: Dengue
Keywords: dengue virus, immunity, hemorrhagic fever, Philippines
MeSH Terms: conditions — Dengue; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Dengue is a common disease and a major health concern in the Philippines. Dengue is caused by a virus transmitted from the bite of an infected mosquito. The purpose of this study is to understand why some infants remain well or have a mild illness, and why other infants become very sick from this virus. Studies have shown that the mother's immune response to dengue can play a role in the infant's immune response and affect whether or not the infant becomes sick. This study will enroll up to 10,000 healthy infants 6-14 weeks old and their mothers in San Pablo City. At the first study visit, information about the mother and birth will be collected and blood samples will be taken from the mother and infant. The infant will have blood drawn at all 3 study visits. The infants will be followed until the age of 16 months. The information obtained from this study may help in the development and future testing of a safe and effective dengue vaccine.

DETAILED DESCRIPTION:
This is a prospective natural history study to define the levels of maternally-acquired neutralizing antibody (Ab) and other correlates of immunity that may protect against the development of dengue hemorrhagic fever in infants. Approximately 10,000 mother-infant pairs will be enrolled to achieve a continuous study cohort of approximately 4,000 children less than 16 months of age. Children leave the study when they reach 16 months of age and are replaced by new participants at 6-14 weeks of age. The investigators will recruit study participants among 3rd trimester pregnant women receiving pre-natal care and women with newborns receiving post-natal care in San Pablo City. The first aim of this study is to define levels of serotype-specific neutralizing Abs associated with protective immunity against symptomatic dengue virus (DV). Neutralizing Ab titers in blood samples collected from Filipino infants before DV infection, and predicted neutralizing Ab titers at the time of illness, will be correlated with disease severity rankings and peak viremia levels. Neutralizing Ab titers at which infants developed symptomatic dengue will be determined. The second aim will be to delineate risk factors contributing to the pathogenesis of dengue hemorrhagic fever (DHF) in infants. From pre-illness blood samples, the association of Ab neutralizing capacity or enhancement of infection with DHF will be measured while controlling for other potential covariates. The covariates will include measures representing viral load and infant host immune responses. The third aim will be to strengthen the capacity for diagnosis and research on dengue in the Philippines. A collaborative and international consortium has been formed to advance dengue research in the Philippines. The research will generate vital data for the effective testing of dengue vaccines and future public health vaccination campaigns throughout the region. This study will enroll up to 10,000 healthy infants 6-14 weeks old and their mothers in San Pablo City. The infants will be followed until the age of 16 months. Mothers and infants will enter the study when the infant is between the ages of 6-14 weeks. At the 1st study visit, data on the mother and the birth will be collected and blood samples will be collected from the mother and infant. The infant will have blood drawn at all 3 study visits. The 2nd study visit will take place when the infant is between the ages of 4-6 months. At this time, data on infant health will be obtained. In all infants, an anticoagulated blood sample will be collected for plasma and PBMC isolation. At age 15-16 months, 250 infants per year will be selected to return for a 3rd study visit. The 250 infants will be randomly selected from those without prior symptomatic dengue and whose study visits 2 and 3 span a significant portion of the peak DV transmission season (June-October). Data on infant health will be obtained and an anticoagulated blood sample for plasma will be collected. Surveillance for DV infections will occur year round and throughout the entire period of an infant's study participation (ages 6 weeks-16 months). Study personnel will screen infants in the study who present with acute febrile illnesses. Those infants will have history and clinical data abstracted, and an acute illness blood sample (serum) taken for dengue diagnostic testing. A convalescent blood sample (serum) will also be taken 10-14 days later. The primary outcome measured will be the identification of DV infection and the classification of disease severity. The secondary outcome measured will be the estimation of peak viremia levels.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born to mother residing in San Pablo Health District
2. Planned residence in San Pablo Health District for at least 1 year
3. Age 6-14 weeks*
4. Informed consent
5. General good health * Except on study initiation, when over the first 5 months of Year 1 (est. Feb-June 2006), infants between the ages of 6-24 weeks will be allowed to enter the study.

Exclusion Criteria:

1. Infant born with congenital medical disorder
2. Mother known to be HIV seropositive

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20000
Dates: Start 2006-09; Study Completion 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Tropical Medicine, City of Muntinlupa, Philippines

REFERENCES:
- [Derived] Libraty DH, Acosta LP, Tallo V, Segubre-Mercado E, Bautista A, Potts JA, Jarman RG, Yoon IK, Gibbons RV, Brion JD, Capeding RZ. A prospective nested case-control study of Dengue in infants: rethinking and refining the antibody-dependent enhancement dengue hemorrhagic fever model. PLoS Med. 2009 Oct;6(10):e1000171. doi: 10.1371/journal.pmed.1000171. Epub 2009 Oct 27. PMID 19859541